CLINICAL TRIAL: NCT01620749
Title: A Phase 0 Exploratory Microdosing Study of 6-18fluoro-N-[2-(Diethylamino)Ethyl]Pyridine-3-carboxamide (18F MEL050) Using PET/CT in Patients With Metastatic Melanoma
Brief Title: Of 18F MEL050 Using PET/CT in Metastatic Melanoma
Acronym: MEL050
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cooperative Research Centre for Biomedical Imaging Development (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10/11
Record Dates: First submitted 2012-05-27; First posted 2012-06-15 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: Metastatic Melanoma
Keywords: melanoma metastatic diagnosis
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MEL050 (Experimental)
  Interventions: Radiation: 18F MEL050

INTERVENTIONS:
Radiation: 18F MEL050 — Diagnostic intervention to establish the safety and biodistribution of MEL050 in participants with melanoma.

SUMMARY:
The purpose of this study is to investigate the safety and potential effectiveness of the imaging compound 18F MEL050 for finding sites of melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained prior to any protocol-specific procedures
* Male and female patients with histologically confirmed melanoma
* At least one site of metastatic disease, as demonstrated on the pre-study 18F FDG PET/CT scan performed as part of routine clinical care
* Age >/= 18 years
* Life expectancy >/=3 months
* ECOG performance score of 0-2

Exclusion Criteria:

* Pregnant or breastfeeding females
* Systemic anti-melanoma therapy within the 2 weeks prior to the pre-study 18F FDG PET/CT scan until after the 18F MEL050 PET/CT scan
* Patients whose clinical care may be compromised because of the delay resulting from performance of the 18F MEL050 PET/CT scan
* Patients whose only metastatic lesion is in the Central Nervous System
* Patients with urinary incontinence or patients who cannot comfortably hold their urine for more than 90 minutes
* Any serious medical condition which the investigator feels may interfere with the procedures or evaluations of the study
* Patients unwilling or unable to comply with protocol and patients with a history of non compliance or inability to grant informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-06; Primary Completion 2012-03 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Safety of 18F MEL050 administration as measured by occurrence of adverse clinical, biochemical or haematological events following 18F MEL050 administration. | Up to 28 days following 18F MEL050 administration (+/- 7 days)

SECONDARY OUTCOMES:
Percentage of injected 18F MEL050 dose in organs of interest. | 10, 30, 60 and 120 minutes post 18F MEL050 administration
Percentage of unmetabolized 18F MEL050 in plasma and urine after radiotracer administration. | 60, 120 and 180 minutes post 18F MEL050 administration.
Absorbed organ doses and whole body dose expressed as milliSv/200MBq administered dose. | 10, 30, 60 and 120 minutes post 18F MEL050 administration

CONTACTS AND LOCATIONS:
Overall Officials: Grant McArthur, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (1):
- Peter MacCallum Cancer Centre, East Melbourne, Victoria, Australia